CLINICAL TRIAL: NCT04374968
Title: Use of Blood Flow Restriction (BFR) Therapy in Peri-operative Rehabilitation Following Anterior Cruciate Ligament Tear
Brief Title: Use of Blood Flow Restriction Therapy Following ACL Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Joseph Tramer, Resident Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13080
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Anterior Cruciate Ligament Tear; Knee Injuries; Sport Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial with a treatment and control group
Who Masked: Outcomes Assessor
Masking Description: Participant and investigator will be aware of treatment arm allocation. Outcomes will be assessed in a masked fashion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- BFR Treatment (Experimental): Patients will be recruited following ACL tear and medical screening for history of DVT/PE. Patients allocated to the BFR intervention group will undergo physical therapy with the use of a blood flow restriction cuff. Rehabilitation will consist of a structured home exercise program prior to surgery. We will instruct patients on how to perform home BFR and test them in the office to ensure competence. Following surgery patients will immediately be started in physical therapy. Therapy will consist of a structured program progressing from range of motion, to strength training and then functional tests. Both arms will use the same protocol with the only difference being use of BFR.
  Interventions: Device: Blood flood restriction cuff
- Control (No Intervention): The control arm will undergo the same pre and post operative physical therapy as the BFR group. They will undergo a structure home therapy program prior to surgery and an outpatient physical therapy program under the guidance of a therapist following surgery.

INTERVENTIONS:
Device: Blood flood restriction cuff — Blood flow restriction cuffs will be used as an augment to physical therapy
  Arms: BFR Treatment

SUMMARY:
Evaluating the use of peri-operative blood flow restriction therapy surrounding anterior cruciate ligament tear

DETAILED DESCRIPTION:
The purpose of this study is to examine the effect of utilizing blood flow restriction (BFR) therapy both before and after anterior cruciate ligament reconstruction (ACLR) following a tear. BFR has been proposed to work by restricting arterial inflow leading to an oxygen depleted environment and the ability to induce muscle adaption at lower maximum repetition via reactive hyperemia. Muscle atrophy occurs following ACL tear and reconstruction. Thus, physical therapy is used in the peri-operative period to regain strength with the ultimate goal of returning to activity.

The goal of this investigation is to determine if using BFR during perioperative therapy would lead to increased and expedited strength gains. Additionally we would like to determine if BFR helps patients to pass the standard rehabilitative functional tests and return to play sooner. We will also look at patient reported outcomes metrics and pain scores to determine if BFR has a significant impact on the patient experience surrounding ACL tear and reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* ACL tear undergoing reconstruction

Exclusion Criteria:

* History of pulmonary embolism
* History of deep vein thrombosis
* Family history of PE/DVT
* Hypercoaguable disorder
* Multiligamentous knee injury
* Neurovascular injury
* Peripheral vascular disease
* Unable to complete physical therapy
* Unable to tolerate blood flow restriction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Quadriceps Strength | Three months
  Quadriceps strength via handheld dynamometer

SECONDARY OUTCOMES:
Quadriceps Strength | six months
  Quadriceps strength via handheld dynamometer
Knee range of motion | three months
  Knee range of motion via goniometer
Knee range of motion | six months
  Knee range of motion via goniometer
Patient reported outcome measurement information system | Three months
  Patient reported outcomes measurement information system score on patient physical function, scale 0-100 with higher scores better
Patient reported outcomes measurement information system | Six months
  Patient reported outcomes measurement information system score on patient physical function, scale 0-100 with higher scores better
international knee documentation committee questionnaire | three months
  international knee documentation committee questionnaire, scale 0-100 with higher scores better
international knee documentation committee questionnaire | six months
  international knee documentation committee questionnaire, scale 0-100 with higher scores better
Pain scores | three months
  Visual analog scale pain scores, scale 0-10 higher is more pain
Pain scores | six months
  Visual analog scale pain scores, scale 0-10 higher is more pain

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, West Bloomfield, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okoroha KR, Tramer JS, Khalil LS, Jildeh TR, Abbas MJ, Buckley PJ, Lindell C, Moutzouros V. Effects of a Perioperative Blood Flow Restriction Therapy Program on Early Quadriceps Strength and Patient-Reported Outcomes After Anterior Cruciate Ligament Reconstruction. Orthop J Sports Med. 2023 Nov 27;11(11):23259671231209694. doi: 10.1177/23259671231209694. eCollection 2023 Nov. PMID 38035216